CLINICAL TRIAL: NCT07169253
Title: Comparison of GAP, ILD-GAP, and CPI in Idiopathic Pulmonary Fibrosis (IPF) and Hypersensitivity Pneumonitis (HP)
Brief Title: Prognostic Score Comparison in IPF and HP
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ERDOGAN CETINKAYA, Prof. Dr., Saglik Bilimleri Universitesi
Other Study IDs: ILDPrognostic-Scores
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: IPF; Fibrotic Lung Disease; Hypersensitivity Pneumonitis; Interstitial Lung Disease (ILD)
Keywords: Idiopathic Pulmonary Fibrosis; Hypersensitivity Pneumonitis; GAP; ILD-GAP; CPI
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IPF: The demographic data, symptom duration, clinical and laboratory findings, radiological images, BAL results, and histopathological diagnoses of patients diagnosed with IPF were evaluated according to the 2018 ATS/ERS/JRS/ALAT Clinical Practice Guideline for the Diagnosis of IPF and included in the IPF group.
  Interventions: Other: GAP Index; Other: ILD-GAP Index; Other: Composite Physiologic Index (CPI)
- Fibrotic HP: Patients diagnosed with fibrotic HP were classified according to the 2020 ATS/JRS/ALAT Clinical Practice Guideline for the Diagnosis of Hypersensitivity Pneumonitis in Adults.
  Interventions: Other: GAP Index; Other: ILD-GAP Index; Other: Composite Physiologic Index (CPI)
- Non-fibrotic HP: Patients diagnosed with non-fibrotic HP were classified according to the 2020 ATS/JRS/ALAT Clinical Practice Guideline for the Diagnosis of Hypersensitivity Pneumonitis in Adults.
  Interventions: Other: GAP Index; Other: ILD-GAP Index; Other: Composite Physiologic Index (CPI)

INTERVENTIONS:
Other: GAP Index — For each patient in the IPF, fibrotic HP, and non-fibrotic HP groups, the GAP index was calculated based on age, gender, FVC, and DLCO values. According to the GAP index, patients were classified as Stage 1 (0-3 points), Stage 2 (4-5 points), and Stage 3 (6-8 points).
Other: ILD-GAP Index — In addition to the GAP parameters, the index was calculated to include the ILD subtype as well.
Other: Composite Physiologic Index (CPI) — The CPI (Composite Physiologic Index) was calculated using the following formula:
  CPI = 91 - (0.65 × %DLCO) - (0.53 × %FVC) + (0.34 × %FEV1).
  DLCO: Diffusing Capacity of the Lung for Carbon Monoxide FVC: Forced Vital Capacity FEV₁: Forced Expiratory Volume in One Second

SUMMARY:
The goal of this retrospective observational study is to evaluate and compare the prognostic value of GAP, ILD-GAP, and CPI scoring systems in patients diagnosed with interstitial lung diseases (ILDs), specifically Idiopathic Pulmonary Fibrosis (IPF), fibrotic Hypersensitivity Pneumonitis, and non-fibrotic Hypersensitivity Pneumonitis.

The main questions it aims to answer are:

* Can GAP, ILD-GAP, and CPI scores accurately predict prognosis in IPF, fibrotic HP, and non-fibrotic HP patients?
* Are there differences in prognostic performance of these models across different ILD subtypes?

Researchers will compare the prognostic utility of GAP, ILD-GAP, and CPI scores between IPF, fibrotic HP, and non-fibrotic HP groups to see if one scoring system offers superior predictive power.

Participants:

* Adults aged ≥18 years
* Diagnosed between October 2011 and October 2021 at the University of Health Sciences Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital
* 143 patients in total (IPF: 45, fibrotic HP: 26, non-fibrotic HP: 72)

Participants' data will include:

* Clinical and demographic characteristics
* Symptom duration
* Radiologic imaging findings
* Pulmonary function test (PFT) results
* Bronchoalveolar lavage (BAL) findings
* Histopathological diagnoses

Scoring systems will be calculated using standardized formulas as follows:

* GAP (Gender, Age, Physiology)
* ILD-GAP (modified GAP for CTD-ILDs)
* CPI (Composite Physiologic Index = 91 - [0.65 × %DLCO] - [0.53 × %FVC] + [0.34 × %FEV1])

DETAILED DESCRIPTION:
This is a retrospective observational study designed to evaluate and compare the prognostic performance of three widely used scoring systems-Gender-Age-Physiology (GAP) Index, Interstitial Lung Disease-GAP (ILD-GAP) Index, and Composite Physiologic Index (CPI)-in patients diagnosed with interstitial lung diseases (ILDs). The study focuses specifically on three ILD subtypes: Idiopathic Pulmonary Fibrosis (IPF), fibrotic Hypersensitivity Pneumonitis (HP), and non-fibrotic HP.

The primary objective is to determine whether GAP, ILD-GAP, and CPI scores can accurately predict overall survival across these patient groups. A secondary aim is to compare the prognostic performance of the scoring systems to explore whether one model provides superior predictive value in specific ILD subtypes.

The study cohort includes adult patients (≥18 years) who were diagnosed between October 2011 and October 2021 at the University of Health Sciences Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital. A total of 143 patients were identified and included: 45 patients with IPF, 26 with fibrotic HP, and 72 with non-fibrotic HP.

Data collected for each patient include clinical and demographic characteristics, duration of symptoms, high-resolution computed tomography (HRCT) findings, pulmonary function test (PFT) results, bronchoalveolar lavage (BAL) findings, and histopathological diagnoses where available. The final diagnosis in each case was established through multidisciplinary team (MDT) discussions and/or histopathological confirmation.

The scoring systems were calculated using standardized formulas:

GAP Index: based on gender, age, and physiology (FVC % predicted, DLCO % predicted).

ILD-GAP Index: a modification of the GAP model for use in connective tissue disease-associated and other ILDs.

CPI (Composite Physiologic Index): calculated as 91 - (0.65 × %DLCO) - (0.53 × %FVC) + (0.34 × %FEV1).

By applying these validated prognostic models to a real-world ILD cohort, the study aims to provide insights into their relative accuracy, clinical utility, and potential limitations. Findings are expected to contribute to more precise prognostic assessment and risk stratification in patients with fibrotic and non-fibrotic ILDs.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients diagnosed with IPF based on clinical features, laboratory findings, thoracic HRCT results, and/or histopathological confirmation, as determined by a multidisciplinary team discussion.
* 40 patients diagnosed with Fibrotic Hypersensitivity Pneumonitis based on clinical features, laboratory findings, and thoracic HRCT results, confirmed in a multidisciplinary team discussion.
* 40 patients diagnosed with Non-Fibrotic Hypersensitivity Pneumonitis based on clinical features, laboratory findings, and thoracic HRCT results, confirmed in a multidisciplinary team discussion.
* Male and female patients over 18 years of age.

Exclusion Criteria:

* Patients under 18 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Chronic Hypersensitivity Pneumonitis (fibrotic/non-fibrotic) and Idiopathic Pulmonary Fibrosis (IPF) by multidisciplinary discussion between October 2011 and October 2021 at the University of Health Sciences Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Prognostic performance of the Gender-Age-Physiology (GAP) Index, Interstitial Lung Disease-GAP (ILD-GAP) Index, and Composite Physiologic Index (CPI) in predicting overall survival | Using data collected between October 2011 and October 2021
  Prognostic performance of GAP, ILD-GAP, and CPI scoring systems in predicting overall survival among patients with Idiopathic Pulmonary Fibrosis (IPF), fibrotic Hypersensitivity Pneumonitis, and non-fibrotic Hypersensitivity Pneumonitis.

SECONDARY OUTCOMES:
Association between clinical parameters and survival across ILD subgroups | Using data collected between October 2011 and October 2021
  Evaluation of the relationship between patient age, gender, presence of comorbidities, and symptom profiles and overall survival in IPF, fibrotic HP, and non-fibrotic HP groups using log-rank tests and Cox regression.
Impact of CPI score increase on mortality risk | Using data collected between October 2011 and October 2021
  Assessment of the association between each 1-unit increase in Composite Physiologic Index (CPI) and the risk of mortality using Cox proportional hazards regression.
Effect of GAP stage, gender, and CTD status on survival | Using data collected between October 2011 and October 2021
  Stratified survival analysis to investigate whether GAP stage (I-III), female gender, and absence of connective tissue disease are associated with longer survival, using Kaplan-Meier curves and multivariate Cox models.
Comparison of prognostic performance (AUC) of GAP, ILD-GAP, and CPI across ILD subtypes | At baseline scoring and during follow-up (using data collected between October 2011 and October 2021)
  Receiver Operating Characteristic (ROC) analysis to compare the discriminative ability of GAP, ILD-GAP, and CPI scores in predicting mortality. AUC values were reported for each model across IPF, fibrotic HP, and non-fibrotic HP subgroups.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)